CLINICAL TRIAL: NCT03133442
Title: Effect of Vestibular Stimulation on Sleep in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SOMNOMAT V4
Record Dates: First submitted 2017-04-05; First posted 2017-04-28 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: The study has a two-by-two cross-over design. Participants spend two consecutive baseline nights (without stimulation) and two consecutive movement nights (with stimulation) in the laboratory. The order of baseline and movement nights is randomized.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of the participants is impossible, as the stimulation is easy to perceive and cannot be confused with a baseline night. Therefore, participants are informed about the character of the night (max. 5 minutes) before the moment of lights off. For safety reasons the experimenter that is present is also aware of the condition.
  However, data is stored in a coded way, so that during data analysis the experimenter is not aware of the condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline Nights (No Intervention): No vestibular stimulation is applied. However, the sound of the moving bed will be played back to the participant at the right sound intensity level.
- Movement Nights (Experimental): Vestibular stimulation, in the form of gentle rocking movements, is provided using the Somnomat V4 rocking bed. Stimulation is provided for the entire 7 hours of the night from lights off to lights on. The stimulation frequency is in the range of 0.1-0.3 Hz, with an amplitude in the range of 0.05 to 0.1m
  Interventions: Device: Somnomat V4

INTERVENTIONS:
Device: Somnomat V4 — Vestibular stimulation is provided using an innervated bed platform. This robotic device consists of a standard single bed, mounted on a moving mechanism. It was developed and produced by the ETH Zürich and approved for use in this study by Swissmedic.
  Arms: Movement Nights

SUMMARY:
Vestibular stimulation might be beneficial for sleep. Previous research demonstrated that lateral rocking movements can facilitate the transition from wake to sleep during an afternoon nap. However, the relationship between rocking movements and sleep is poorly understood to date. Furthermore, studies looking at the effects of rocking on sleep have not yet been performed in an elderly population. Due to age related changes in sleep, people often experience a decrease in sleep efficiency and sleep quality later in life. Therefore, it is particularly this population that could benefit from a possible enhancement in sleep efficiency and sleep quality. In order to assess the effect of vestibular stimulation on sleep and sleep-dependant memory, measurements of two nights with stimulation will be compared to two baseline nights. The primary outcomes are changes in sleep onset, sleep architecture and power density spectra of the EEG due to vestibular stimulation. Secondary endpoints are sleep dependent changes in memory, the proximal-distal temperature gradient, cardiorespiratory variables and dream content.

ELIGIBILITY:
Inclusion Criteria:

* Right handed
* Between 60 and 75 years of age

Exclusion Criteria:

* Diseases or lesions of the nervous system (acute or residual included neurological and psychiatric diseases)
* BMI < 19 or > 30 kg/m2
* Medication known to influence sleep [56]
* Cognitive Impairment (MoCA score < 26)
* Drug use and abuse
* Nicotine use (e.g. smoking)
* > 10 alcoholic drinks per week
* > 5 drinks or foods containing caffeine per day
* History of sleep disorder (Insomnia, sleep apnea (apnea-hypopnea index >5), nocturnal myoclonus (>5 periodic leg movements per hour of sleep))
* Irregular sleep-wake rhythm (e.g. shift working)
* Travelling across time zones less than 1 month ago
* Naps longer than 1h
* Sleep on an average night <6 hours or >8 hours
* Skin allergies or very sensitive skin
* Diseases of the vestibular system
* Signs of motion sickness based on questionnaire

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-12 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Polysomnography | 4 nights of 7 hours each
  Difference in sleep parameters between the second of two nights with intervention and the second of two nights without intervention, as recorded using polysomnography. The sleep stages will be scored visually on a 20-s epoch basis according to standard criteria [53]. This will allow us to compare sleep architecture of the participants in the two conditions, as well as a possible consecutive nights effect in the two movement nights. Parameters of specific interest are sleep onset latency, total sleep time, time spent in N1, N2 and N3 stages of NREM sleep and time spent in REM sleep.
  Furthermore, the EEG power density spectra will be analysed. Power in specific frequency bands will be calculated based on spectral analysis, the amount and density of sleep spindles and slow waves will be determined.

SECONDARY OUTCOMES:
Memory performance | Recall moment in evening and morning (4 nights)
  Difference in declarative memory performance between the second of two nights with intervention and the second of two nights without intervention. During each experimental night a word-pair recall task will be performed 1h before going to bed and half an hour after waking up. To assess declarative memory performance improvement, we will determine the difference between immediate and delayed recall. Word-pair recall tasks are suitable to determine declarative memory performance in the context of sleep, as they are sensitive to effects of sleep.
Skin temperature | 4 nights of 7 hours each
  The distal-proximal temperature gradient will be calculated, based on skin temperature measured using sensors placed on the chest and hands, to look for a relationship with sleep onset latency.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riener, Prof., Principal Investigator — University of Zurich
Locations (1):
- Sensory Motor Systems Lab, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No